CLINICAL TRIAL: NCT04455490
Title: Clinical Effect of Endoscopic Surgery for Delayed Wound Healing After Achilles Tendon Suture
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2019492
Record Dates: First submitted 2020-06-25; First posted 2020-07-02 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-07

CONDITIONS: Wound Healing
Keywords: Achilles tendon suture; Delayed wound healing; Endoscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Delayed wound healing: Patients with delayed wound healing after Achilles tendon suture who were treated at Peking University Third Hospital
  Interventions: Other: Self-control

INTERVENTIONS:
Other: Self-control — We compared relevant scores of patients before and after surgery

SUMMARY:
This study proposes endoscopic surgery for delayed wound healing after Achilles tendon suture which is a brand new treatment，and retrospectively analyzed the clinical data of 4 cases treated with this treatment. The analysis results of the clinical efficacy of the method can serve as a reference for clinical and surgical decision-making and prognosis assessment.

DETAILED DESCRIPTION:
Background: Delayed wound healing is a kind of postoperative complication of Achilles tendon suture. Conventional surgical approach is open surgery in order to clean the wound, which requires multiple dressing changes and involves a longer recovery period. We recently developed arthroscopic surgery for delayed wound healing after Achilles tendon suture. This therapy may be an alternative approach to open surgery.

Purposes: In this paper we evaluate the long-term efficacy of endoscopic surgery for delayed wound healing after Achilles tendon suture.

Patients and Methods: Clinical data of 4 patients with delayed wound healing after Achilles tendon suture who underwent endoscopic surgery from April 2008 to October 2017 at our institute were retrospectively analyzed. There were 3 males and 1 females with age of 39-60 years, the follow-up period was 8-43 months). All the patients had unilateral tendon rupture with 3 cases on the left and 1 cases on the right. Scores on Visual analogue scale(VAS) and the American Orthopaedic Foot and Ankle Society (AOFAS) Ankle-Hindfoot Scale were used. The postoperative outcome was evaluated on the basis of Victorian Institute of Sport Assessment-Achilles score and Achilles tendon total rupture score (ATRS).

ELIGIBILITY:
Inclusion Criteria:

* The diagnostic criteria for delayed wound healing after Achilles tendon suture are met, namely the presence of skin necrosis, wound nonunion, or delayed wound healing.

Exclusion Criteria:

* The expected healing time of wounds with regular dressing changes is <2 weeks.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 4 patients with delayed healing after Achilles tendon suture surgery who were treated at our institution, in the period from April 2008 to July 2019. The patients were 3 men and 1 woman, aged 39 to 60 years. Among them, 3 had surgery on the left Achilles tendon and 1 had surgery on the right Achilles tendon. The time from the first operation (Achilles tendon suture) to foreign body reaction ranged from 1 month to 5 months.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2020-03-18 (Actual); Primary Completion 2020-04-18 (Actual); Study Completion 2020-05-18 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 8 months to 4 years after the surgery
  Use Visual Analog Scale(VAS) to evaluate the pain recovery of patients who received endoscopic surgery. VAS ranges from 0 to 10, higher scores mean a worse outcome.
American Orthopaedic Foot and Ankle Society Ankle-Hindfoot Score | 8 months to 4 years after the surgery
  Use American Orthopaedic Foot and Ankle Society Ankle-Hindfoot Score(AOFAS) to evaluate the function recovery of patients who received endoscopic surgery. AOFAS ranges from 0 to 100, higher scores mean a better outcome.
Victorian Institute of Sport Assessment-Achilles | 8 months to 4 years after the surgery
  Use Victorian Institute of Sport Assessment-Achilles(VISA-A) to evaluate the pain and movement recovery of patients who received endoscopic surgery. VISA-A ranges from 0 to 100, higher scores mean a better outcome.
Achilles tendon total rupture score | 8 months to 4 years after the surgery
  Use Achilles tendon total rupture score(ATRS) to evaluate the function and movement recovery of patients who received endoscopic surgery. VISA-A ranges from 0 to 100, higher scores mean a better outcome.
Tegner knee motion score | 8 months to 4 years after the surgery
  Use Tegner knee motion score to evaluate the sports ability of patients who received endoscopic surgery. Tegner knee motion score ranges from 0 to 10, higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No